CLINICAL TRIAL: NCT02410720
Title: The Effectiveness of a Customized Mobile Application in Colonoscopy Preparation: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Customized Mobile Application in Colonoscopy Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ala'a Sharara, Professor of Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IM.AS1.35
Record Dates: First submitted 2013-07-10; First posted 2015-04-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Colonoscopy Preparation
Keywords: Colonoscopy Preparation; Polyethylene Glycols; Mobile application; Software; Compliance; Patient Compliance; Adherence
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Instruction leaflet (Active Comparator): Patients will receive the Picoprep solution with an instruction leaflet of how to use it and the dietary modifications needed
  Interventions: Other: Instruction leaflet; Other: Explanation of paper and application instructions; Other: Picoprep solution
- Mobile App (Experimental): Patients will receive Picoprep solution with an instruction leaflet + Picoprep Mobile App which will be downloaded to their smartphones that has the same information plus a reminder utility
  Interventions: Other: Instruction leaflet; Other: Mobile App; Other: Explanation of paper and application instructions; Other: Picoprep solution

INTERVENTIONS:
Other: Instruction leaflet — Patients will receive the Picoprep solution with an instruction leaflet of how to use it and the dietary modifications needed
Other: Mobile App — Patients will receive Picoprep solution with an instruction leaflet + Picoprep Mobile App which will be downloaded to their smartphones that has the same information plus a reminder utility
  Arms: Mobile App
Other: Explanation of paper and application instructions — The research fellow will explain instructions to patients
Other: Picoprep solution

SUMMARY:
Colonoscopy is the preferred procedure to investigate any large-bowel disease in adults and children. In addition, colonoscopy is the current gold standard for colorectal cancer screening due to its high diagnostic capabilities and its unique feature that permits sampling and removal of pathology. For optimal performance and visualization of details, however, an adequate bowel preparation is essential. Inadequate bowel preparation is associated with cancelled procedures, prolonged procedure time, incomplete examination, increased cost and possibly complications, physician frustration and patient anxiety, but most importantly serving to impede colorectal cancer screening and surveillance.

A good bowel preparation would need a solution with a reasonable volume, acceptable taste, minimal diet restrictions, and easy to follow instructions; and would also need patients' adherence to the instructions and diet restrictions. Noncompliance of patients to the diet restrictions, the starting day of diet, the timing of drinking the solution, and other instructions play an important role in rendering the colon preparation inadequate.

Aim: The investigators aim, at assessing the influence of having a reminder mobile application on the compliance and adherence to instructions and diet and consequently on the quality of colon preparation.

Hypothesis: The investigators' hypothesis is that patients having a customized mobile App reminding them systematically about instruction and time of intake of the preparation will have a better adherence to the prep protocol and likely on the quality preparation than those given written and verbal instructions in clinic.

DETAILED DESCRIPTION:
This is a randomized controlled trial that will include patients undergoing elective colonoscopy at the American University of Beirut Medical Center. Patients will be randomized into one of two study arms using a computer generated randomization list. 160 patients will be enrolled in total. All patients will be instructed by the study coordinator on the importance of adherence to the protocol in the leaflet emphasizing its importance to the colonoscopy quality. In addition, patients in Arm 2 will be given information about the application features. The application will have push notifications to inform patient on time of start of dietary changes, type of diet, time of preparing the solution, time of drinking the solution, reminder of their appointment, etc. All patients will then be interviewed by the research coordinator to evaluate the adherence to the assigned diet and compliance with the prep protocol as the main outcome and the ease of the application and the patient's attitude towards having such application as secondary outcomes. Based on the results of similar studies that assessed the use of software system to improve compliance, the investigators' sample size was a calculated assuming similar results. Calculations showed that 78 patients per arm will be enough to attain significance. The number 80 was chosen as attrition is presumed to be low. As for the statistical analysis, SPSS version 20.0 will be used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Elective outpatient colonoscopy
* Consent to the study
* Owning a smartphone

Exclusion Criteria:

* Pregnant or lactating women
* Age less than 18 years
* Known Inflammatory bowel disease
* Significant gastroparesis
* Gastric outlet obstruction
* Ileus
* Known or suspected bowel obstruction or perforation
* Phenylketonuria
* Toxic colitis or megacolon
* Having a stoma
* Compromised swallowing reflex or mental status
* Psychiatric disease or known or suspected poor compliance
* Severe chronic renal failure (creatinine clearance <30 mL/minute)
* Severe congestive heart failure (New York Heart Association [NYHA] class III or IV)
* Dehydration
* Laxative use or dependency
* Chronic constipation (<3 spontaneous bm/week)
* Uncontrolled hypertension (systolic blood pressure ≥170 mm Hg, diastolic blood pressure ≥100 mm Hg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Quality of the preparation using the modified Aronshick scale | Directly after the Colonoscopy
  During every colonoscopy a blinded interventionalist will assess the quality of the preparation using the modified Aronshick scale
Questionnaire for adherence to the assigned diet | 30 minutes before the Colonoscopy
  The research coordinator will ask the patients specific questions to assess their adherence to the assigned diet ( first and second dietary changes)
Questionnaire for compliance with the prep protocol | 30 minutes before the Colonoscopy
  The research coordinator will ask the patients specific questions to assess their compliance with the prep protocol

SECONDARY OUTCOMES:
Patient satisfaction with the written instructions and mobile application using a visual analogue scale | 30 minutes before the Colonoscopy
  Patient satisfaction will be assessed using a visual analogue scale
Questionnaire for ease of use of the mobile App | 30 minutes before the Colonoscopy
  Patients will be asked about the ease of use of the mobile App
Questionnaire for patient willingness to take the same preparation in the future if needed | 30 minutes before the Colonoscopy
  Patients will be asked about their willingness to take the same preparation in the future if needed

CONTACTS AND LOCATIONS:
Overall Officials: Ala' I Sharara, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Sharara AI, Chalhoub JM, Beydoun M, Shayto RH, Chehab H, Harb AH, Mourad FH, Sarkis FS. A Customized Mobile Application in Colonoscopy Preparation: A Randomized Controlled Trial. Clin Transl Gastroenterol. 2017 Jan 5;8(1):e211. doi: 10.1038/ctg.2016.65. PMID 28055031